CLINICAL TRIAL: NCT01537445
Title: MR-Evaluation of Renal Function-After-Pancreas-transplantation
Acronym: MERFAP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Per Liss, Associate professor, Uppsala University
Other Study IDs: MERFAP-2012
Record Dates: First submitted 2012-02-13; First posted 2012-02-23 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes; Renal Failure; Pancreas Transplantation
Keywords: Diabetes Mellitus; Pancreas; Renal failure; Transplantation
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with pancreastransplantation: All patients undergoing pancreas transplantation.

SUMMARY:
The purpose of this study is to evaluate the beneficial effect of pancreas transplantation for long term kidney function in patients undergoing single-pancreas transplantation.

DETAILED DESCRIPTION:
Renal failure in patients who have performed a pancreas transplantation is a hazard for the outcome for these patients. The beneficial effect of pancreas transplantation for renal function is not clear. It is of major importance to early find patients who develops a decrease in renal function and start treatment early and closely monitor these patients in order to avoid further deteriorating renal function. In order to achieve this, there is a need for a easy, fast and sensitive method to evaluate renal function. In this study the investigators plan to use the non-invasive MR to evaluate changes in renal function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus
* Patients undergoing a pancreas transplantation

Exclusion Criteria:

* Patients undergoing a pancreas transplantation and a renal transplantation at the same time.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Kidney function | Within 3 years
  Improvements in kidney function (GFR) and proteinuria after pancreas transplantation.

SECONDARY OUTCOMES:
Kidney hemodynamics and oxygenation | Within 3 years
  Improvements in renal blood flow and kidney tissue oxygenation after pancreas transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Per Liss, MD, PhD., Study Director — Uppsala University, Uppsala, Sweden
Locations (1):
- University Hospital, Uppsala, Uppsala County, Sweden